CLINICAL TRIAL: NCT06123065
Title: Yoga for Warriors: A Pilot Study of Feasibility and Efficacy of A Yoga Intervention for Veterans With Comorbid Chronic Pain and PTSD
Brief Title: Feasibility and Efficacy of A Yoga Intervention for Comorbid Chronic Pain and PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hunter Holmes Mcguire Veteran Affairs Medical Center (U.S. Federal Agency)
Collaborators: Virginia Commonwealth University (Other); McGuire Research Institute (Other)
Responsible Party: Principal Investigator, Suzzette M. Chopin, PhD, Study PI, Hunter Holmes Mcguire Veteran Affairs Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1572859
Record Dates: First submitted 2023-10-30; First posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: PTSD; Chronic Pain
Keywords: Yoga; Virtual Intervention
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Chronic Pain | interventions — Yoga

STUDY DESIGN:
Intervention Model Description: Delayed cross-over design, with a Waitlist control. This study was a quasi-randomization to Active or Waitlist and Waitlist individuals were then moved to the Active group after assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Immediately enrolled into Yoga intervention. Completed orientation and baseline measures then began 8-week yoga group intervention.
  Interventions: Behavioral: Yoga
- Waitlist (Other): Delayed Intervention. Waitlist individuals attended orientation and completed baseline measures. After completion of re-assessment of measures 8 weeks later, then enrolled into Active arm.
  Interventions: Behavioral: Yoga

INTERVENTIONS:
Behavioral: Yoga — 8 week Yoga for chronic pain and PTSD group intervention, conducted virtually
  Other Names: Complementary and Alternative Intervention

SUMMARY:
The goal of this pilot quasi-randomized study is test the feasibility, acceptability, and initial efficacy of Yoga for Warriors treatment program for comorbid chronic pain and PTSD, conducted virtually through the Richmond Veterans Affairs Medical Center (RICVAMC).

the main questions it aims to answer are:

1. Whether a virtual intervention for chronic pain and PTSD is feasible and acceptable for veterans.
2. Using a wait-list control group design, to determine preliminary efficacy of the intervention.
3. Examine follow-up data to determine if benefits are maintained over time.

DETAILED DESCRIPTION:
The study will be a pilot quasi-randomized controlled design comparing the 8-session Yoga for Warriors program, conducted via a web-based platform, utilizing a wait-list control, with wait-list participants being enrolled in subsequent groups. Measures of treatment satisfaction will be given and rates of initiation following screening and drop-out will be measured. A battery of assessments will be given at baseline (group introduction), at mid-point (around session 4), and following completion of the group. To determine maintenance effects, select assessments and re-administration of the study assessment battery will be conducted 3 months post-completion.

Potentially interested participants will be screened for eligibility. Screening for eligibility will occur over the phone and those who are interested in participating and willing to engage in the online format and who meet inclusion criteria based on study staff screening will go through the informed consent process over the phone or virtually. Collection of informed consent from participants will not include written documentation of informed consent given the fully virtual nature of this study during the coronavirus pandemic (COVID-19) restrictions (waiver of documentation of consent has been submitted). Paperless recording of willingness to participate will take place, with no written documentation of consent to participate. Participants will attend an initial online orientation session (prior to the first yoga session), either in a group format or individually, where they will be provided information on the group, will be randomized into the treatment group or to the wait-list control group. To attend the orientation session and all yoga sessions, participants will be emailed the specific, secured link to the online platform. Participants will complete the measures over the phone with the study coordinator. This will be an 8 week (+1 orientation session) group conducted remotely, online, with additional self-report measures completed mid-treatment, post-treatment, and at follow-up, in the same manner as described above.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic pain (defined as pain for > 3 months) in the electronic medical record and a score of 50 or more on the Pain Disability Questionnaire (PDQ)
* Probable PTSD defined as being above the clinical threshold on the PTSD Checklist for DSM-5 (PCL-5), sum score at or above 25
* Able to stand up from sitting on the floor without assistance
* Able to ambulate community distances without an assistive device
* Intact sensation in lower extremities below knees
* Medical clearance by primary care provider
* Access to a computer/laptop/ipad with internet and video capability.

Exclusion Criteria:

* Fall risk
* Pregnancy
* Joint replacement within the past 12 months
* Active alcohol/other substance abuse or dependence (unless actively engaged in treatment)
* Current psychotic disorder or hospitalization with psychotic symptoms in past 3 months
* Active (past 3 months) suicidal or homicidal ideation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
PTSD Checklist for Diagnostic and Statistic Manual for Mental Disorders 5 (DSM-5) | past week; assessed at baseline, mid-treatment (after week 4), post-treatment (after week 8), 3 month follow up
  Assess current symptoms of PTSD in line with DSM-5 criteria (20 items)
Pain Disability Questionnaire | past week; assessed at baseline, mid-treatment (after week 4), post-treatment (after week 8), 3 month follow up; Items rated on 1 to 10-point scale; higher scores indicate worse outcome
  Assesses self report of impact of pain in functioning (15 items)
Pain Catastrophizing Scale | current; past week; assessed at baseline, mid-treatment (after week 4), post-treatment (after week 8), 3 month follow up; Items rated 0 to 4; higher scores indicate worse outcomes
  Assesses self report of thoughts and worries related to chronic pain (13 items)

SECONDARY OUTCOMES:
Client Satisfaction Questionnaire-8 (CSQ-8) | Time in intervention; Assessed at post-treatment (8 weeks); Items rated 1 to 4; higher scores indicate better outcomes
  Th CSQ is an 8-item measure assesses general intervention satisfaction
Patient Health Questionnaire-9 (PHQ-9) | Past 2 weeks; assessed at baseline and post-treatment (8 weeks); Items rated 0 to 3; higher scores indicate worse outcomes
  The PHQ-9 assesses depression severity
Generalized Anxiety Disorder 7-Item Scale (GAD-7) | Past 2 weeks; assessed at baseline and post-treatment (8 weeks); Items rated 0 to 3; higher scores indicate worse outcomes
  The GAD-7 measures anxiety experienced
Patient Reported Outcome Measurement Information System (PROMIS) Short Form Anger | Past 7 days; assessed at baseline and post-treatment (8 weeks); Items rated 1 to 5; raw scores converted to T scores; higher scores mean worse outcomes
  Assesses emotional distress and anger (5 items)
Patient Reported Outcome Measurement Information System (PROMIS) Short Form Social Roles | Past 7 days; assessed at baseline and post-treatment; (8 weeks); Items rated 1 to 5; raw scores converted to T scores; higher scores mean better outcomes
  Assesses ability to participate in social roles and activities
Tampa Scale for Kinesiophobia (TSK-11) | Current; assessed at baseline, mid-treatment (4 weeks), post-treatment (8 weeks), 3 month follow up; Items rated 1 to 4; higher scores indicate worse outcomes
  The TSK-11 is an 11-item scale used to measure general perceptions of pain interference
Quality of Life Enjoyment and Satisfaction Questionnaire -- Short Form (LES-Q-SF) | past week; assessed at baseline, post-treatment (8 weeks), 3 month follow up; Items rated 1 to 5; higher scores indicate better outcomes
  The Q-LES-Q-SF is a 16-item scale used to measure quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Suzzette Chopin, Ph.D., Principal Investigator — Richmond Veteran Affairs Medical Center
Locations (1):
- Richmond Veterans Affairs Medical Center, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Fully de-identified participant level data and aggregate data (all collected IPD) will be made available to qualified researchers who contact the Study PI per the Institutional Review Board's approved data management and sharing plan.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Starting 6 months following publication of primary dataset. Data will remain available for up to 10 years.
Access Criteria: Qualified researchers (i.e., based on degree and institutional support) who request de-identified data from study PI (listed as corresponding author) following publication of primary paper. Relevant data dictionaries and analytic scripts may also be shared through encrypted email or file-sharing programs. PI/corresponding author will review requests and make final approval decisions for data sharing.

REFERENCES:
- [Background] Chopin SM, Sheerin CM, Meyer BL. Yoga for warriors: An intervention for veterans with comorbid chronic pain and PTSD. Psychol Trauma. 2020 Nov;12(8):888-896. doi: 10.1037/tra0000649. Epub 2020 Jul 23. PMID 32700935
- [Derived] Chopin SM, Zaur AJ, Fountain C, Claros Nunez A, Sheerin CM. Feasibility of a Virtual Adaptation of a Yoga Intervention for Veterans with Chronic Pain and Posttraumatic Stress Disorder. J Integr Complement Med. 2025 Jan;31(1):92-99. doi: 10.1089/jicm.2024.0512. Epub 2024 Sep 10. PMID 39253832